CLINICAL TRIAL: NCT00942526
Title: The Correlation of Oral Anti-Infective Agent With Anastomotic Leakage in Reconstruction Surgery for Esophageal Cancer
Brief Title: Oral Anti-Infective Agent for Esophageal Anastomotic Leakage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Pei-Ming Huang, Department of Surgery, National Taiwan University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 200806035R
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Anastomotic Leakage
Keywords: esophageal cancer; anastomotic leakage; Prevention of anastomotic leakage after esophageal surgery
MeSH Terms: conditions — Anastomotic Leak; Esophageal Neoplasms | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): no intervention with perioperative oral anti-infective agent or water for gargling
- 2 (Sham Comparator): perioperative gargling with water
  Interventions: Other: Water
- 3 (Experimental): perioperative oral gargling with oral anti-infective agent for seven days
  Interventions: Drug: Mycostatin oral suspension

INTERVENTIONS:
Drug: Mycostatin oral suspension — peroperative Mycostatin oral suspension ( 0.1MU/cc, 24cc/bt; 5cc qid)for 7 days
  Arms: 3
Other: Water — perioperative gargling with water
  Arms: 2

SUMMARY:
Anastomotic leakage is still to be a major cause of considerable morbidity and mortality after esophagectomy and gastric pull up for esophageal carcinoma. Risk factor analyses of anastomotic leakage, including blood supply, graft tension, and comorbidity, have been performed, but few studies have produced strategies that have improved operative results. This study will be performed to identify prognostic variables that might be used to develop a strategy for optimizing outcomes after esophagogastrectomy.

DETAILED DESCRIPTION:
Goal:

The effect of oral hygiene on the occurrence of esophagogastric anastomotic leakage has not yet been studied for along time. We will use a random cohort study model and investigate the effect of perioperative oral anti-infective gargle agent on the esophagogastric anastomotic wound healing.

Method:

1. Design:

   One hundred and twenty patients are divided into 3 groups and each group has 40 esophageal patients. Minimization stratified randomization will be applied. Oral anti-infective gargling agent, Mycostatin oral suspension, will be employed for one week before operation. The first groups will be treated without oral gargle agent; the second groups will be treated with gargling water; and the third groups will be treated with anti-infective gargling agent.

   An end-to-side two-layer esophagogastric anastomosis will be constructed using interrupted sutures with metallic staple through cervical wound. On the other hand, the anastomotic leakage rates in different groups will be investigated.
2. Data Collection and Statistic Analysis:

The records of all patients, various biologic parameters, and the management of leakage are analyzed. Thirty-day morbidity and mortality are determined, and stepwise multivariable logistic regression analysis assesses the effect of preoperative and postoperative variables on anastomotic leakage. Time variation of starting oral feeding and hospital stay are compared using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* carcinoma of the esophagus, operable stage I to III

Exclusion Criteria:

* patients who were inoperable,
* patients who had obvious impaired blood supply of gastric substitutes, and
* patients who had non-cervical esophagogastrostomy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
all cause anastomotic leakage | two years

SECONDARY OUTCOMES:
Time variation of starting oral feeding and hospital stay | two years

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ming Huang, MD, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Liu K, Zhang GC, Cai ZJ. Avoiding anastomotic leakage following esophagogastrostomy. J Thorac Cardiovasc Surg. 1983 Jul;86(1):142-5. PMID 6865459
- [Background] Roy-Choudhury SH, Nicholson AA, Wedgwood KR, Mannion RA, Sedman PC, Royston CM, Breen DJ. Symptomatic malignant gastroesophageal anastomotic leak: management with covered metallic esophageal stents. AJR Am J Roentgenol. 2001 Jan;176(1):161-5. doi: 10.2214/ajr.176.1.1760161. PMID 11133560
- [Background] Bardini R, Asolati M, Ruol A, Bonavina L, Baseggio S, Peracchia A. Anastomosis. World J Surg. 1994 May-Jun;18(3):373-8. doi: 10.1007/BF00316817. PMID 8091778
- [Background] Peracchia A, Bardini R, Ruol A, Asolati M, Scibetta D. Esophagovisceral anastomotic leak. A prospective statistical study of predisposing factors. J Thorac Cardiovasc Surg. 1988 Apr;95(4):685-91. PMID 3280882
- [Background] Dewar L, Gelfand G, Finley RJ, Evans K, Inculet R, Nelems B. Factors affecting cervical anastomotic leak and stricture formation following esophagogastrectomy and gastric tube interposition. Am J Surg. 1992 May;163(5):484-9. doi: 10.1016/0002-9610(92)90393-6. PMID 1575303
- [Background] Patil PK, Patel SG, Mistry RC, Deshpande RK, Desai PB. Cancer of the esophagus: esophagogastric anastomotic leak--a retrospective study of predisposing factors. J Surg Oncol. 1992 Mar;49(3):163-7. doi: 10.1002/jso.2930490307. PMID 1548890
- See also: National Taiwan University Hospital (NTUH) Research Ethics Committee (REC) — http://www.ntuh.gov.tw/RECO